CLINICAL TRIAL: NCT04716088
Title: Usefulness of Rapid Antigen Testing for SARS-CoV-2 Among Healthcare Workers to Prevent Spread of COVID-19 in the Hospital: a Pilot Study
Brief Title: Rapid Antigen Testing for SARS-CoV-2 Among Healthcare Workers to Prevent Spread of COVID-19
Status: Completed | Type: Observational
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Collaborators: Insitute of Microbiology and Immunology, Faculty of Medicine, University of Ljubljana (Unknown)
Responsible Party: Sponsor
Other Study IDs: RADT for COVID-19 Golnik
Record Dates: First submitted 2021-01-15; First posted 2021-01-20 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: SARS-CoV-2 Rapid Antigen Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Rapid antigen test for SARS CoV2 — Defining diagnostic performance of repeated testing regimen in hospital setting

SUMMARY:
Physicians, nurses and hospital attendants currently working at the University Clinic of Respiratory and Allergic Diseases Golnik were invited to participate in the pilot study. Nasopharyngeal swabs were obtained three times per week for two consecutive weeks and tested with a point-of-care rapid antigen test and reverse transcription polymerase chain reaction (RT-PCR). In addition, serum samples were obtained at the beginning of the study and 2 weeks after last swab was obtained in order to evaluate the serological status of participating health care workers.

DETAILED DESCRIPTION:
Health care workers (HCW) currently working at the University Clinic of Respiratory and Allergic Diseases Golnik were invited to enroll in the pilot study. HCW directly involved in COVID-19 patient care and those who had a previous laboratory confirmed SARS-CoV-2 infection were not eligible for inclusion in the study. For each participating HCW, nasopharyngeal swabs were obtained. Swabs were collected on Mondays, Wednesdays and Fridays for two consecutive weeks with a maximum of six samplings per person scheduled.

Swabs were inserted into universal transport medium (UTM) and tested with SARS-CoV-2 Rapid Antigen test (Roche Diagnostics GmbH, Mannheim, Germany), in accordance with the manufacturer's instructions. Briefly, samples were thoroughly vortexed and 350 μL of UTM were mixed with the extraction buffer included in the testing kit. Three drops of the mixture were applied to the specimen well of the lateral flow test device and results were visually read after a 15 min incubation at room temperature.

Nasopharyngeal swab samples were subsequently tested for the presence of SARS-CoV-2 RNA without intermitting freeze-thaw cycle. Viral RNA was isolated from the specimens using the QIAamp Viral RNA Mini Kit (QIAGEN GmbH, Hilden, Germany). PCR amplification was set up on CFX96 Touch Real-Time PCR Detection System (Bio-Rad Laboratories - Dubai Branch, Dubai, United Arab Emirates) and a commercially available PCR kit Allplex™2019-nCoV (Seegene, Seoul, South Korea) was used. Allplex™2019-nCoV assay enables simultaneous detection and identification of three target genes, specific for SARS-CoV-2 (e.g. the E, RdRp, and N gene). Samples were considered positive for SARS-CoV-2 only if all three targeted genes were amplified.

In addition, serum samples were collected at the beginning of the study and 14 days after the last nasopharyngeal swab was obtained. The presence of antibodies against SARS-CoV-2 were evaluated using IDK anti-SARS-CoV-2 IgM and IgG ELISA Kit (Immundiagnostik AG, Bensheim, Germany), following manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* health care worker

Exclusion Criteria:

* previous known COVID 19 infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physicians, nurses and hospital attendants currently working at the University Clinic of Respiratory and Allergic Diseases Golnik were invited to enroll in the pilot study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
SARS CoV2 infection | 14 days
  positive rapid antigen test for SARS CoV2

CONTACTS AND LOCATIONS:
Overall Officials: Mihaela Zidarn, MD PhD, Principal Investigator — Klinika Golnik
Locations (1):
- Universitiy Clinic for respiratory and allergic diseases, Golnik, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided
IPD are available on request from PI.

REFERENCES:
- [Derived] Jakobsen KK, Jensen JS, Todsen T, Tolsgaard MG, Kirkby N, Lippert F, Vangsted AM, Martel CJ, Klokker M, von Buchwald C. Accuracy and cost description of rapid antigen test compared with reverse transcriptase-polymerase chain reaction for SARS-CoV-2 detection. Dan Med J. 2021 Jun 14;68(7):A03210217. PMID 34169830
- [Derived] Sterbenc A, Tomic V, Bidovec Stojkovic U, Vrankar K, Rozman A, Zidarn M. Usefulness of rapid antigen testing for SARS-CoV-2 screening of healthcare workers: a pilot study. Clin Exp Med. 2022 Feb;22(1):157-160. doi: 10.1007/s10238-021-00722-y. Epub 2021 May 22. PMID 34021827